CLINICAL TRIAL: NCT00002422
Title: A Phase I/II, Open-Label Study of the Safety, Tolerance, Pharmacokinetics, Drug-Interaction and Anti-HIV Activity of Intramuscularly Administered Alpha-Epi-Br (HE2000) in HIV-Infected Patients on Salvage Therapy
Brief Title: A Study on the Safety and Anti-HIV Activity of HE2000 in HIV-Infected Patients on Salvage Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Harbor Therapeutics (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 303A; HE2000-005
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2009-06-25 (Estimated); Status verified 2002-04

CONDITIONS: HIV Infections
Keywords: Injections, Intramuscular; Drug Interactions; Salvage Therapy; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — 16alpha-bromo-3beta-hydroxy-5alpha-androstan-17-one

INTERVENTIONS:
Drug: HE2000

SUMMARY:
The purpose of this study is to see if it is safe and effective to give HE2000, an experimental anti-HIV drug, to HIV-infected patients on salvage therapy (emergency treatment used when a patient has not responded to standard therapy).

HE2000 is a hormone that is suspected to make it more difficult for HIV to live in cells.

DETAILED DESCRIPTION:
HE2000 is a synthetic steroid hormone that, when tested in the laboratory, had anti-viral activity against wild-type and drug-resistant variants of HIV. HE2000 works through a natural biochemical mechanism in cells to make them less able to support viral infection.

There are 4 treatment groups of increasing doses of HE2000; each group consists of 2 parts (Part A and B). Part A is a single administration of HE2000 injected intramuscularly, and Part B is 5 consecutive daily intramuscular injections of HE2000. Patients receive the same dosage throughout Parts A and B of the study. Patients are asked to return to the clinic periodically for blood sample collection. Patients may remain at the hospital overnight for pharmacokinetic evaluation. Drug safety, tolerance, efficacy, and pharmacokinetics are measured. Samples from treatment Group 4 are analyzed for specific cell function.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are at least 18 years old.
* Are HIV-positive.
* Have been on their current anti-HIV drug combination for at least 30 days prior to the screening visit.
* Are currently failing at least their second anti-HIV drug treatment.
* Are not responding to their current anti-HIV treatment, have failed at least 1 anti-HIV combination, and do not have many options for treatment (Groups 3 and 4 only).
* Are willing to not make any changes in their anti-HIV treatment until at least Day 50 during the study.
* Have a CD4 count of at least 100 cells/mm3 at study entry.
* Have a viral load (level of HIV in the body) between 5,000 and 250,000 copies/ml at study entry.
* Agree to use barrier methods of birth control (e.g., condoms) during the study.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have hepatitis B or C.
* Have been treated for cancer within 4 weeks prior to study entry, or will need to be treated during the study. (Patients with Kaposi's sarcoma are eligible but must not have received any treatment within 4 weeks before study entry or require treatment during the study.)
* Have received certain medications including those affecting the immune system.
* Are pregnant or breast-feeding.
* Have an active, serious infection, including opportunistic (AIDS-defining) infection that requires treatment during the study or during the 2 weeks prior to study entry.
* Have a condition or are receiving therapy that would prevent them from completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - ViRx Inc, Palm Springs, California
  - Veterans Affairs Palo Alto Health Care Ctr, Palo Alto, California
  - Quest Clinical Research, San Francisco, California
  - Northwestern Univ Med School, Chicago, Illinois
  - St Vincents Hosp / Clinical Research Program, New York, New York
  - Plaza Med Ctr, Houston, Texas